CLINICAL TRIAL: NCT01961531
Title: BrUOG 291: FIVE FRACTION PARTIAL BREAST IRRADIATION USING NON-INVASIVE IMAGE-GUIDED BREAST BRACHYTHERAPY (NIBB)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brown University (Other)
Collaborators: Watson Clinic Cancer Center (Other); Cancer Treatment Centers of America (Other); University of California, San Diego (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 291
Record Dates: First submitted 2013-10-10; First posted 2013-10-11 (Estimated); Results first posted 2020-08-25 (Actual); Last update posted 2022-03-04 (Actual); Status verified 2022-02

CONDITIONS: Breast Cancer
Keywords: DCIS; IDC; Invasive breast carcinoma
MeSH Terms: conditions — Breast Neoplasms; Carcinoma, Intraductal, Noninfiltrating

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Accuboost APBI (Experimental): 28Gy delivered in 5 daily fractions
  Interventions: Device: Accuboost APBI

INTERVENTIONS:
Device: Accuboost APBI — 28Gy delivered in 5 daily fractions

SUMMARY:
To evaluate safety of 5 fraction accelerated partial brest irradiation in more convenient 5 fraction schedule.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the rate of early and intermediate toxicity related to accelerated partial breast irradiation (APBI) delivered in a more convenient 5 fraction schedule using non-invasive image-guided breast brachytherapy (NIBB) (AccuBoost System) in women with resected, early stage breast cancer.

Non-invasive image-guided breast brachytherapy (NIBB), using advanced image-guided radiation technology, has the potential to eliminate the disadvantages of the conventional APBI techniques. NIBB facilitates non-invasive partial breast irradiation without the use of catheters or implants. Yet by using breast immobilization and precise image-guidance, it reduces non-target breast tissue within the irradiated field compared with other non-invasive APBI techniques such as 3D-CRT. This has made NIBB an attractive approach to deliver APBI.

We hypothesize that NIBB delivered in 5 treatments will be a more convenient, safe and effective modality to deliver partial breast irradiation.

Anticipated advantages of NIBB protocol treatment include:

* Convenient treatment schedule
* Short course can allow for increased patient access to treatment
* Non-invasive approach
* Increased accuracy with precise targeting of lumpectomy cavity using advanced imaging
* Reduced irradiation of non-target breast tissue
* Reduced skin toxicity
* No heart or lung radiation exposure
* Reduced late skin or breast toxicity
* High rate of good or excellent cosmetic outcome
* High rate of ipsilateral breast tumor control comparable to other APBI techniques

ELIGIBILITY:
Inclusion Criteria:

1. A confirmed histological diagnosis of invasive breast carcinoma or DCIS;
2. Age greater or equal to 50 years old;
3. Life expectancy > 6 months;
4. Treated by breast conserving surgery
5. Pathologic lymph node negative, which includes (pN0 i-, i+);

   Patients, who are at very low risk for sentinel node involvement and sentinel node biopsy is not performed, are eligible if the treating investigator documents clinically lymph node negative (cN0). These patients include:
   * DCIS
   * Microinvasion only
   * Pure tubular or mucinous histology
   * Patients ≥ 70yo with T1a-T1c; estrogen receptor +
6. Pathologic tumor size

   1. less than or equal to 2 cm for invasive disease;
   2. less than or equal to 3 cm for DCIS;
7. Estrogen receptor positive if invasive disease (DCIS can be ER negative)
8. Negative surgical margins greater than or equal to 2 mm. A margin of <2mm is acceptable if at natural boundary, i.e. skin or pectoralis fascia.
9. No lymphovascular invasion;
10. ECOG performance status of 0-2 (Appendix 1);
11. Informed consent signed.

Exclusion Criteria:

1. Known BRCA 1/2 Mutation; (BRCA 1 and 2 testing is not required)
2. Active lupus or scleraderma;
3. Pregnancy;
4. Psychiatric or addictive disorder that would preclude attending follow-up;
5. Neoadjuvant chemotherapy (adjuvant chemotherapy is permitted);
6. Suspicious remaining microcalcification on post-surgery mammogram (unless biopsy proven benign);
7. pN+ on axillary dissection or in the sentinel lymph node biopsy (N0i+ are considered node negative and are not excluded);
8. Multicentric disease;
9. Paget's disease of the nipple;
10. Breast Implants
11. Distant metastases;
12. Lumpectomy cavity not well visualized on AccuBoost imaging;
13. Lumpectomy cavity with 1cm margin (CTV/PTV) not adequately encompassed by any available applicator.
14. Breast separation with compression > 8cm at time of simulation.

Min Age: 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2014-07-24 (Actual); Primary Completion 2016-10-26 (Actual); Study Completion 2021-11-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jaroslaw Hepel, M.D., Principal Investigator — Brown University
Locations (3):
- United States (3):
  - UCSD Moores Cancer Center, La Jolla, California
  - Watson Cancer Center, Lakeland, Florida
  - Rhode Island Hospital, Providence, Rhode Island

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Accuboost APBI
Started | 40
Completed | 40
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Accuboost APBI
Number analyzed (Participants) | 40
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 14
  >=65 years | 26
Age, Continuous [Mean (Full Range); unit: years] | 67.45 [50 to 89]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 0
  Unknown or Not Reported | 40
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 39
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 40

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Any Toxicity Related to the Radiation Treatment
Description: Any toxicity related to the radiation treatment will be scored and graded using National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) v3.0.
Time Frame: during treatment, 2 and 6 weeks post treatment and then every 6 months for up to 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Accuboost APBI
Number analyzed (Participants) | 40
Participants | 40

2. Secondary Outcome: Number of Participants With Ipsilateral Breast Local Recurrence
Time Frame: annually for 2 years post treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Accuboost APBI
Number analyzed (Participants) | 40
Participants | 2

ADVERSE EVENTS:
Time Frame: Data was collected from signing of ICF until 5 years post treatment.
Arm/Group | Accuboost APBI
Serious Adverse Events (participants affected / at risk) | 0/40
Other Adverse Events (participants affected / at risk) | 36/40
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Accuboost APBI (N=40)
Discomfort (General disorders) | 27
Acute Skin Reaction (Skin and subcutaneous tissue disorders) | 32
Skin Induration/Fibrosis (Skin and subcutaneous tissue disorders) | 8
Fatigue (General disorders) | 19
Hyperpigmentation (Skin and subcutaneous tissue disorders) | 7
Breast Soreness (Reproductive system and breast disorders) | 1
Seroma (Musculoskeletal and connective tissue disorders) | 2
Edema (General disorders) | 1
Shoulder Pain (General disorders) | 1
Contralateral Breast Infection (Infections and infestations) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 2
Breast Volume/Hypoplasia (Reproductive system and breast disorders) | 11
Fibrosis-cosmesis (Musculoskeletal and connective tissue disorders) | 3
Telangiectasia (Skin and subcutaneous tissue disorders) | 13
Breast Tenderness (Reproductive system and breast disorders) | 1
Breast Pain (Reproductive system and breast disorders) | 5
Skin Atrophy (Skin and subcutaneous tissue disorders) | 3
Hypopigmentation (Skin and subcutaneous tissue disorders) | 1
Folliculitis (Infections and infestations) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No